CLINICAL TRIAL: NCT04067349
Title: Physical Recovery After Laparoscopic vs. Open Liver Resection - a Pilot Trial
Brief Title: Physical Recovery After Laparoscopic vs. Open Liver Resection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Klaus Kaczirek, Clinical Professor, Medical University of Vienna
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1829/2016)
Record Dates: First submitted 2019-08-21; First posted 2019-08-26 (Actual); Last update posted 2019-08-26 (Actual); Status verified 2019-08

CONDITIONS: Postoperative Complications; Liver Diseases; Physical Stress; Surgery
Keywords: laparoscopic; minimal invasive; physical recovery; liver surgery
MeSH Terms: conditions — Postoperative Complications; Liver Diseases | interventions — Ergometry

STUDY DESIGN:
Intervention Model Description: non-randomized cohort study, 2 parallel groups
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- laparoscopic liver resection (Active Comparator): Patients undergoing laparoscopic liver resection
  Interventions: Other: Ergometry
- open liver resection (Active Comparator): Patients undergoing open liver resection
  Interventions: Other: Ergometry

INTERVENTIONS:
Other: Ergometry — Patients underwent a preoperative ergometry to assess their physical fitness prior to their planned liver resection.
  Bicycle stress testing was performed preoperatively and 1 and 6 months postoperatively.

SUMMARY:
The role of laparoscopic liver surgery with respect to clinical outcome remains unclear.

DETAILED DESCRIPTION:
The role of laparoscopic liver surgery with respect to clinical outcome remains unclear. The investigators hypothesized that laparoscopic liver resection (LLR) is associated with better postoperative recovery than open liver resection (OLR).

Twenty-one patients who underwent LR were included in this study (11 OLR (52.4%) and 10 LLR (47.6%), respectively). Postoperative recovery was measured by bicycle stress testing at months 1 and 6 after surgery and compared to preoperative stress testing. Standardized performance for bicycle stress testing was calculated based on age, sex, height and weight. Postoperative recovery was compared between groups as change of performance (%).

ELIGIBILITY:
Inclusion Criteria:

* all patients undergoing liver resection (open vs. laparoscopic)
* all patients willing participate and gave written informed consent

Exclusion Criteria:

* pregnancy
* significant traumatic injury within 30 days prior to study enrolment
* inability or unwillingness to comply to the protocol or to perform bicycle ergometry

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-04-06 (Actual); Primary Completion 2018-08-08 (Actual); Study Completion 2019-04-14 (Actual)

PRIMARY OUTCOMES:
Overall change in performance | 1, 6 months
  The change in performance after 1 and 6 months postoperatively in comparison to preoperative ergometry.

SECONDARY OUTCOMES:
Postoperative Complications | 1 months
  Secondary endpoints included postoperative complications (wound healing, liver failure, adverse events)
Liver resection and effect on postoperative fitness | 2 years
  patients were divided into two groups ( major (>2 segments) vs. minor (≤2segments) liver resection) and postoperative performance was evaluated
length of stay | 1 month
  Length of postoperative hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Kaczirek, MD, Study Chair — Medical University of Vienna, Department of Surgery
Locations (1):
- Medical University of Vienna, Department of Surgery, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No